CLINICAL TRIAL: NCT00829374
Title: CONCERT: A Phase 3 Multicenter, Randomized, Placebo-Controlled, Double-Blind Twelve-Month Safety and Efficacy Study Evaluating Dimebon in Patients With Mild-to-Moderate Alzheimer's Disease on Donepezil
Brief Title: Safety and Efficacy Study Evaluating Dimebon in Patients With Mild to Moderate Alzheimer's Disease on Donepezil
Acronym: CONCERT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medivation, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIM18
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; clinical trial; mitochondria; memory loss; neurodegenerative disease; dementia; investigational drug
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders; Neurodegenerative Diseases; Dementia | interventions — latrepirdine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Dimebon, 5 mg orally three times daily
  Interventions: Drug: Dimebon
- 2 (Experimental): Dimebon, 20 mg orally three times daily
  Interventions: Drug: Dimebon
- 3 (Placebo Comparator): Placebo orally three times daily
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Dimebon — 5 mg orally three times daily
  Arms: 1
Drug: Dimebon — 20 mg orally three times daily
  Arms: 2
Drug: Placebo comparator — Placebo orally three times daily
  Arms: 3

SUMMARY:
The purpose of this study is to determine if Dimebon is safe and effective in patients with mild to moderate Alzheimer's disease on Donepezil.

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-moderate Alzheimer's disease (AD)
* Probable AD (Diagnostic Statistical Manual of Mental Disorders-IV-Text Revision (DSM-IV-TR))
* Mini-Mental State Examination (MMSE) score between 12 and 24, inclusive
* Stable on donepezil for at least 6 months

Exclusion Criteria:

* Other causes of dementia
* Major structural brain disease
* Unstable medical condition or significant hepatic or renal disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1003 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | Week 52
Alzheimer's Disease Assessment Scale - Cognitive Subscale | Week 52

SECONDARY OUTCOMES:
Clinician's Interview Based Impression of Change, plus caregiver input (CIBIC-plus) | Week 52
Neuropsychiatric Inventory (NPI) | Week 52
Resource Utilization in Dementia Lite (RUD lite) | Week 52
Euro Quality of Life 5 (EQ-5D) | Week 52

CONTACTS AND LOCATIONS:
Locations (101):
- United States (52):
  - Phoenix, Arizona
  - Sun City, Arizona
  - Tucson, Arizona
  - Costa Mesa, California
  - Encino, California
  - Escondido, California
  - Fresno, California
  - Garden Grove, California
  - La Jolla, California
  - Los Alamitos, California
  - Los Angeles, California
  - Martinez, California
  - Newport, California
  - Paramount, California
  - Pasadena, California
  - San Diego, California
  - San Francisco, California
  - Boulder, Colorado
  - Denver, Colorado
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Deerfield Beach, Florida
  - Delray Beach, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Eaton, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Las Vegas, Nevada
  - Mount Arlington, New Jersey
  - Princeton, New Jersey
  - Albany, New York
  - Cedarhurst, New York
  - New York, New York
  - Rochester, New York
  - Durham, North Carolina
  - Beachwood, Ohio
  - Toledo, Ohio
  - Jenkintown, Pennsylvania
  - Norristown, Pennsylvania
  - Providence, Rhode Island
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Seattle, Washington
  - Middleton, Wisconsin
- Australia (7):
  - Newcastle, New South Wales
  - Sydney, New South Wales
  - Brisbane, Queensland
  - Adelaide, South Australia
  - Geelong, Victoria
  - Melbourne, Victoria
  - Perth, Western Australia
- Belgium (3):
  - Antwerp
  - Leuven
  - Sint-Truiden
- Finland (3):
  - Kuppio
  - Oulu
  - Turku
- France (6):
  - Bordeaux
  - Concert
  - Lille
  - Montpellier
  - Nice
  - Toulouse
- Germany (6):
  - Berlin
  - Bochum
  - Freiburg im Breisgau
  - Hattingen
  - Mannheim
  - Munich
- Italy (5):
  - Brescia
  - Florence
  - Genoa
  - Perugia
  - Rome
- New Zealand (2):
  - Christchurch, Canterbury
  - Auckland
- Sweden (3):
  - Malmo
  - Norrköping
  - Stockholm
- United Kingdom (14):
  - Brentford, Middlesex
  - Rushden, Northhamptonshire
  - Glasgow, Scotland
  - Worthington, West Sussex
  - Bath
  - Blackpool
  - Bradford
  - Greater Manchester
  - London
  - Newcastle upon Tyne
  - Norfolk
  - Oxford
  - Southampton
  - Swindon